CLINICAL TRIAL: NCT04867850
Title: Effect of Behavioral Nudges to Clinicians, Patients, or Both on Serious Illness Conversation Documentation for Patients With Cancer
Brief Title: Effect of Behavioral Nudges on Serious Illness Conversation Documentation
Acronym: SPP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 844816; P50CA244690 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Cancer
Keywords: Cancer; Serious Illness Conversation; Machine Learning; Behavioral Economics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible clinicians and patients will be independently randomized to receive nudges using a 2x2 factorial design.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (Active Comparator): Clinicians and patients will receive no further interventions beyond usual practice. Usual care for clinicians includes a nudge consisting of targeted text messages identifying patients at high risk of predicted 6-month mortality based on a validated machine learning prognostic algorithm.
  Interventions: Other: Usual Care
- Clinician Nudge (Experimental): Clinicians receive a nudge consisting of targeted text messages identifying patients at high risk of predicted 6-month mortality based on a validated machine learning prognostic algorithm as well as performance feedback compared to peers.
  Interventions: Other: Clinician Nudge
- Patient Nudge (Experimental): Patients receive a nudge consisting of a normalizing message prompting patients to complete an electronic questionnaire designed to prime patients towards having an SIC.
  Interventions: Other: Patient Nudge
- Clinician and Patient Nudge (Experimental): Both strategies described above will be used.
  Interventions: Other: Clinician Nudge; Other: Patient Nudge

INTERVENTIONS:
Other: Usual Care — Individual clinicians will receive an automated weekly email detailing a weekly roster of their upcoming repeat-patient visits (Index Visit) with patients at high risk of 6-month mortality as determined by a validated machine learning prognostic algorithm. Clinicians will receive a HIPAA compliant text message on the morning of the appointment reminding them to consider a serious illness conversation with patients on the list.
  Arms: Usual Care
Other: Clinician Nudge — Clinicians will receive the usual care weekly email and text message described above under Usual Care. In addition, embedded in the weekly email, clinicians will receive performance feedback information detailing their documented SICs relative to those documented by peers.
  Arms: Clinician Nudge; Clinician and Patient Nudge
Other: Patient Nudge — Ahead of the Index Visit, high risk patients as identified by the prognostic algorithm will receive a nudge via personal text message and email consisting of a normalizing message prompting patients with a personalized link to a short electronic questionnaire on SIC topics.
  Arms: Clinician and Patient Nudge; Patient Nudge

SUMMARY:
The main purpose of this research study is to evaluate the effectiveness of "nudges" to clinicians, to patients, or to both in increasing Serious Illness Conversation (SIC) documentation; and to identify moderators of implementation effects on SIC documentation. The investigators will employ rapid-cycle approaches to optimize the framing of nudges to clinicians and patients prior to initiating the trial and mixed methods to explore contextual factors and mechanisms.

The investigators will conduct a four-arm pragmatic cluster randomize clinical trial to test the effectiveness of nudges to clinicians, nudges to patients, or nudges to both in increasing the frequency and timeliness of SIC documentation in cancer patients vs. usual care (UC). The investigators hypothesize that each of the implementation strategy arms will significantly increase SIC documentation compared to UC and that the combination of nudges to clinicians and to patients will be the most effective.

DETAILED DESCRIPTION:
Patients with cancer often experience physical and emotional distress, utilize unplanned acute care, and undergo medical interventions that are discordant with their wishes. Given the Covid-19 pandemic, these adverse outcomes are amplified, particularly for racial/ethnic minorities. Serious illness conversations (SICs) that elicit patients' values, goals, and care preferences, particularly early in the disease trajectory, are an evidence-based practice, improve patient mood and quality of life, and are recommended by national guidelines. Preliminary data suggests that SICs among patients with cancer are associated with improved quality of life, increased hospice utilization, and decreased acute care utilization. However, most patients with advanced cancer die without a documented SIC and there are well-documented health disparities in implementation for racial and ethnic minorities. Current strategies to promote SICs, including the multi-component strategies of the Serious Illness Conversation Program, focus primarily on clinician education and have marginally increased the timeliness and frequency of SICs and reduced patient anxiety and depression. While core elements of this program are transferable-such as its structured guide-clinical use remains low. For example, even after training, clinicians at Penn Medicine document SICs for fewer than 5% of patients with advanced cancer. There is critical need to develop, test, and disseminate strategies to improve the frequency of SICs.

Implementation strategies informed by behavioral economics are ideally suited to address this problem, which is fundamentally one of clinician and patient behavior change. Clinician barriers to initiating SICs include optimism bias, or the belief that one's own patient is unlikely to experience a negative event; uncertainty about prognosis and appropriate timing; and fear that bringing up end-of-life issues may be distressing to patients. Patient barriers to SIC initiation include fear of discussing the end of life and beliefs that SICs are not appropriate until late in the course of cancer. While previous studies have tested financial incentives for SIC documentation, little research has evaluated behavioral economics-informed strategies to align both clinicians and patients towards earlier SICs.

By intentionally modifying the way choices are framed, behavioral nudges can lead to desirable changes in clinician behavior while preserving clinician choice. The investigators' preliminary work demonstrates the effectiveness of an implementation strategy focusing on a clinician nudge, consisting of performance feedback and targeted text messages identifying patients at high risk of mortality based on a validated machine learning prognostic algorithm. This strategy led to a threefold increase in SIC documentation for high-risk patients, equitably across racial/ethnic minority subgroups, and is now in routine use across Penn Medicine practice sites. However, clinicians still did not document SICs for over half of patients, illustrating the limitations of a clinician-directed implementation strategy alone.

This study will expand on these preliminary findings to evaluate the synergy between clinician- and patient-directed nudges to increase SIC documentation. The main purpose of this research study is to evaluate the effectiveness of nudges to clinicians, to patients, or to both in increasing Serious Illness Conversation (SIC) documentation; and to identify moderators of implementation effects on SIC documentation. The investigators will employ rapid-cycle approaches to optimize the framing of nudges to clinicians and patients prior to initiating the trial and mixed methods to explore contextual factors and mechanisms. The investigators will conduct a four-arm pragmatic cluster randomize clinical trial to test the effectiveness of nudges to clinicians, nudges to patients, or nudges to both in increasing the frequency and timeliness of SIC documentation in cancer patients vs. usual care (UC).

Rationale for clinician nudge using mortality prediction and peer comparison: Due to optimism bias, clinicians routinely overestimate the life expectancy of patients with advanced cancer and delay SICs until too late in the disease course. In part because of this, clinicians reinforce a social norm that early SICs are not part of routine oncology care. Providing an objective assessment of predicted mortality risk may help counteract optimism bias among clinicians and help them identify patients most likely to benefit from SICs. Moreover, that individuals desire to conform to an approved behavior (an injunctive norm) and the behavior of others (a descriptive norm) may contribute to low observed SIC rates, and may also afford an opportunity for intervention. The investigators expect that periodically reminding clinicians of their own performance on SIC documentation, while providing both an injunctive norm (citing national and institutional guidelines) and a descriptive social norm (displaying the behavior of their best performing peers), will lead clinicians to conform more closely to these norms, as has been shown in studies conducted in other contexts.

Rationale for patient nudge using priming: Priming is a type of nudge that frames information to activate one's self-efficacy and willingness to engage in behavior change. This type of nudge has not previously been evaluated as a tool to promote SICs for patients with cancer. The investigators will test the added impact of a patient nudge designed to prime patients and, in turn, their clinicians to having a SIC.

ELIGIBILITY:
Inclusion Criteria:

Clinician (M.D., P.A., or N.P.) participants must meet the following criteria:

1. Provide care at least 1 clinic session per week for adult (age>18 years) patients with solid, hematologic, or gynecologic malignancies at a participating PennMedicine Implementation Lab site

Patient participants must meet the following criteria:

1. Receive care for a solid, hematologic, or gynecologic malignancy from an eligible provider at a participating PennMedicine Implementation Lab site
2. Have at least one scheduled Return Patient Visit (either in person or via telemedicine) with an eligible PennMedicine provider during the study period

Exclusion Criteria:

Clinicians will be ineligible for *any* of the following reasons:

1. Provide exclusively benign hematology, survivorship, and/or genetics care

Patients will be ineligible for *any* of the following reasons:

1. Previously documented SIC within 6 months
2. Have a non-valid phone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4450 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Takvorian, MD, Principal Investigator — University of Pennsylvania; Ravi Parikh, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takvorian SU, Gabriel P, Wileyto EP, Blumenthal D, Tejada S, Clifton ABW, Asch DA, Buttenheim AM, Rendle KA, Shelton RC, Chaiyachati KH, Fayanju OM, Ware S, Schuchter LM, Kumar P, Salam T, Lieberman A, Ragusano D, Bauer AM, Scott CA, Shulman LN, Schnoll R, Beidas RS, Bekelman JE, Parikh RB. Clinician- and Patient-Directed Communication Strategies for Patients With Cancer at High Mortality Risk: A Cluster Randomized Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2418639. doi: 10.1001/jamanetworkopen.2024.18639. PMID 38949813
- [Derived] Takvorian SU, Bekelman J, Beidas RS, Schnoll R, Clifton ABW, Salam T, Gabriel P, Wileyto EP, Scott CA, Asch DA, Buttenheim AM, Rendle KA, Chaiyachati K, Shelton RC, Ware S, Chivers C, Schuchter LM, Kumar P, Shulman LN, O'Connor N, Lieberman A, Zentgraf K, Parikh RB. Behavioral economic implementation strategies to improve serious illness communication between clinicians and high-risk patients with cancer: protocol for a cluster randomized pragmatic trial. Implement Sci. 2021 Sep 25;16(1):90. doi: 10.1186/s13012-021-01156-6. PMID 34563227

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4,450 patients were included in this study on serious illness conversations (SICs). These patients were seen by 163 clinicians across 65 oncologist-advanced practice provider (APP) clusters. Baseline measures and outcome data were collected for patients only.
Units Other Than Participants: Oncologist-APP Clusters
Period: Overall Study
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Started (Oncologist-APP clusters were randomized to receive either the clinician nudge or usual care. Patients were individually randomized to receive the patient nudge or usual care. Combined, the clinician- and patient-directed nudges lead to four combinations of the presence or absence of nudges.) | 1004; 32 Oncologist-APP Clusters | 1179; 33 Oncologist-APP Clusters | 997; 0 Oncologist-APP Clusters | 1270; 0 Oncologist-APP Clusters
Completed | 1004; 29 Oncologist-APP Clusters | 1179; 31 Oncologist-APP Clusters | 997; 0 Oncologist-APP Clusters | 1270; 0 Oncologist-APP Clusters
Not Completed | 0; 3 Oncologist-APP Clusters | 0; 2 Oncologist-APP Clusters | 0; 0 Oncologist-APP Clusters | 0; 0 Oncologist-APP Clusters

BASELINE CHARACTERISTICS:
Population: Baseline measures, participant counts, and outcome data all correspond to details for patients only. Baseline and outcome data were not collected for clinicians.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge | Total
Number analyzed (Participants) | 1004 | 1179 | 997 | 1270 | 4450
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 74] | 68 [59 to 75] | 67 [58 to 74] | 68 [59 to 75] | 67 [59 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 556 | 594 | 558 | 644 | 2352
  Male | 448 | 585 | 439 | 626 | 2098
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 29 | 28 | 36 | 122
  Not Hispanic or Latino | 975 | 1150 | 969 | 1234 | 4328
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 1 | 4
  Asian | 23 | 28 | 43 | 35 | 129
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 2 | 2 | 7
  Black or African American | 192 | 206 | 176 | 196 | 770
  White | 736 | 873 | 722 | 963 | 3294
  More than one race | 4 | 6 | 10 | 9 | 29
  Unknown or Not Reported | 48 | 62 | 43 | 64 | 217
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1004 | 1179 | 997 | 1270 | 4450
Predicted odds of 180-day mortality (based on a validated machine learning algorithm; 0-1 scale) [Median (Inter-Quartile Range); unit: Avg. predicted probability of mortality] — To be enrolled in this study, patients needed to have been identified as having high six-month mortality risk (>10%). Using a validated machine learning algorithm, risk scores (expressed as the percent chance of dying within six months) were calculated for patients before potentially being added to the study.
  Avg. predicted probability of mortality | .18 [.13 to .30] | .19 [.13 to .33] | .18 [.13 to .32] | .19 [.13 to .33] | .19 [.13 to .32]

OUTCOME MEASURES:

1. Primary Outcome: Number of High Risk Patients With Documentation of a Serious Illness Conversation (SIC)
Description: Measured at the patient level as a binary outcome (yes/no) among high-risk patients based on date of documented note including the SIC template in the Advanced Care Planning (ACP) section of the electronic medical record by any provider
  Outcomes were measured for patients only.
Time Frame: Within 6 months of the Index Visit (baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 1004 | 1179 | 997 | 1270
Participants | 112 | 136 | 115 | 179

2. Secondary Outcome: Number of Patients With SIC Documentation (Out of All Patients, Regardless of Risk Level)
Description: Measured at the patient level as a binary outcome (yes/no) among all cancer patients based on date of documented note including the SIC template in the Advanced Care Planning (ACP) section of the electronic medical record by any provider
  Outcomes were measured for patients only.
Time Frame: Within 6 months of first repeat patient visit during trial period
Population: Data were not collected for this outcome because it reflected a different patient population than the one in this study. The workflow for identifying patients for this trial was based on patients having a risk score (risk of predicted 180-day mortality based on a validated machine-learning prognostic algorithm) exceeding a certain threshold ahead of their clinical appointment, and it was infeasible to track patients with a risk score below this threshold.
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of High Risk Patients With a Palliative Care Referral
Description: Measured at the patient level as a binary outcome (yes/no) among high-risk patients based on presence of a scheduled palliative care appointment
  Outcomes were measured for patients only.
Time Frame: Within 6 months of the Index Visit (baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 1004 | 1179 | 997 | 1270
Participants | 84 | 94 | 81 | 97

4. Secondary Outcome: Number of Decedent High Risk Patients Who Received Aggressive End-Of-Life Care
Description: Measured at the patient level as a binary outcome (yes/no) among high-risk patients who die based on the presence of any of the following three criteria: chemotherapy within 14 days before death, hospitalization within 30 days before death, or admission to hospice 3 days or less before death
  Outcomes were measured for patients only.
Time Frame: Within 6 months of the Index Visit (baseline)
Population: Aggressive End-Of-Life Care was only assessed among the 773 decedents.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
Number analyzed (Participants) | 162 | 227 | 157 | 227
Participants | 76 | 95 | 62 | 97

ADVERSE EVENTS:
Time Frame: For each patient, adverse events were tracked for six months following baseline.
Description: All outcomes and adverse events were tracked for patients only.
Arm/Group | Usual Care | Clinician Nudge | Patient Nudge | Clinician and Patient Nudge
All-Cause Mortality (participants affected / at risk) | 162/1004 | 227/1179 | 157/997 | 227/1270
Serious Adverse Events (participants affected / at risk) | 0/1004 | 0/1179 | 0/997 | 0/1270
Other Adverse Events (participants affected / at risk) | 0/1004 | 0/1179 | 0/997 | 0/1270

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT04867850/Prot_SAP_000.pdf